CLINICAL TRIAL: NCT07144254
Title: Study of Tegavivint, a Transducin Beta-like Protein 1 (TBL1) Inhibitor, With Gemcitabine in Patients With Relapsed or Refractory Osteosarcoma
Brief Title: Tegavivint With Gemcitabine in Patients With Relapsed or Refractory Osteosarcoma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Iterion Therapeutics (Industry)
Responsible Party: Principal Investigator, William T Cash, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00008647
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Osteosarcoma Recurrent; Osteosarcoma in Children; Relapsed Osteosarcoma; Refractory Osteosarcoma
Keywords: Tegavivint; TBL1 inhibitor; Gemcitabine; Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tegavivint with Gemcitabine (Experimental): Subjects can receive treatment with tegavivint and gemcitabine for up to 17 cycles (1 cycle = 21 days). Treatment will be discontinued if there is progressive disease or toxicity requiring treatment discontinuation
  Dose Escalation:
  Dose level 0: Tegavivint = 3(mg/kg) and Gemcitabine 1000 (mg/m2) Dose level 1: Tegavivint = 5(mg/kg) and Gemcitabine 1000 (mg/m2) Dose level 2: Tegavivint = 6.5(mg/kg) and Gemcitabine 1000 (mg/m2)
  Interventions: Drug: Tegavivint; Drug: Gemcitabine

INTERVENTIONS:
Drug: Tegavivint — Tegavivint will be administered second, IV over 4 hours, on days 1, 8, and 15 at the dose level assigned at study entry Cycle length will be 21 days. A cycle may be repeated for a total of 17 cycles, up to a total duration of therapy of approximately 12 months.
Drug: Gemcitabine — Gemcitabine will be administered first, intravenously (IV) over 60 minutes, on days 1 and 8 at a fixed dose of 1000 mg/m2

SUMMARY:
The goal of this clinical trial is to define the maximum tolerated dose (MTD) and/or Recommended phase 2 dose (RP2D) of Tegavivint in combination with Gemcitabine in patients with relapsed or refractory osteosarcoma (OS).

The study will also investigate the toxicities of Tegavivint in combination with gemcitabine in patients with relapsed or refractory OS.

DETAILED DESCRIPTION:
Recurrent osteosarcoma (OS) has a poor prognosis, with 5-year overall survival after relapse ranging from 13% to 45%. There are currently no chemotherapy agents proven to significantly improve survival in relapsed or refractory OS, particularly in patients with unresectable disease, highlighting the need for new treatments.

Tegavivint is a first-in-class small molecule that targets the Wnt/beta-catenin signaling pathway by inhibiting the TBL1-beta-catenin complex, leading to beta-catenin degradation and suppression of oncogenic transcription without affecting its normal cellular functions.

Tegavivint showed potent anti-tumor activity in OS cell lines and mouse models, inhibiting tumor growth and metastasis, including activity against chemoresistant and cancer stem-like cells.

Recent clinical data shows:

Adults: In a Phase 1/2a trial (NCT03459469) with 24 patients, tegavivint at 5 mg/kg (3 weeks on/1 week off) was well tolerated with no dose-limiting toxicities. Most side effects were mild (fatigue, nausea, headache), and serious toxicities common to other Wnt inhibitors were not seen. Tumor shrinkage (>50%) occurred in five patients, with others achieving prolonged stable disease.

Pediatrics: In an ongoing COG Phase 1/2 trial (NCT04851119), tegavivint was tested in 10 patients at 5 and 6.5 mg/kg. No DLTs were observed, and the recommended dose was set at 6.5 mg/kg. Most side effects were grade 1-2; grade ≥3 events were infrequent.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis:

Participants must have had histologic verification of osteosarcoma at original diagnosis or relapse.

* All participants with relapsed or refractory osteosarcoma are eligible, provided they received front-line treatment with a regimen that contained at least 3 of the following agents: methotrexate, doxorubicin, cisplatin, and ifosfamide

  -Disease Status:
* Dose Escalation: Participants must have either measurable or evaluable disease per RECIST.Note: Participants with no evidence of disease on imaging (e.g., following pulmonary metastasectomy) are not eligible during the dose escalation phase.
* Dose Expansion: Participants with measurable or evaluable disease per RECIST and those with no evidence of disease on imaging following pulmonary metastasectomy are eligible during the dose expansion phase.

  -Performance Level: Participants must have a Lansky (≤ 16 years) or Karnofsky (> 16 years) score of ≥ 60, or Eastern Cooperative Oncology Group (ECOG) ≤ 2 Note: Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory to assess the performance score.

  -Prior Therapy: Participants must have fully recovered from the clinically significant acute effects of all prior anti-cancer chemotherapy, immunotherapy, surgery, or radiation therapy before enrollment.
* Myelosuppressive chemotherapy: ≥ 14 days after the last dose.
* Hematopoietic growth factors: ≥ 14 days after a long-acting growth factor (e.g., pegfilgrastim) or ≥ 7 days for a short-acting growth factor. For agents with known delayed adverse events, extend recovery period accordingly.
* Biologic (anti-neoplastic) agent: ≥ 7 days after the last dose. Extend period if adverse events occur beyond 7 days.
* Cellular therapy: ≥ 21 days since last dose (e.g., modified T cells, gamma-delta T cells, natural killer (NK) cells, dendritic cells) with recovery from associated toxicities.
* Interleukins, interferons, and cytokines (excluding hematopoietic growth factors): ≥ 21 days since last dose.
* Antibodies: 7 days or 3 half-lives (whichever is longer), up to 30 days. Toxicity must be resolved to Grade ≤ 1.
* Radiation therapy (XRT):

  * 14 days after local palliative XRT (small port)
  * 150 days after radiation to ≥ 50% of pelvis or bone marrow
  * 6 weeks after substantial bone marrow radiation

Prior use of Nucleoside Analogue (Gemcitabine): Allowed. Investigational agents not otherwise specified: ≥ 30 days since last dose. Surgery: ≥ 2 weeks since last major surgery, including pulmonary metastasectomy (central line placement and core/small open biopsies are excluded)

Organ Function Requirements:

* Adequate Bone Marrow Function Defined As:

  * Peripheral absolute neutrophil count (ANC) ≥ 750/mm3 (0.75x109/L)
  * Platelet count ≥ 75,000/mm3 (75x109/L)
* Adequate Renal Function Defined As: Creatinine clearance or radioisotope GFR ≥ 70 ml/min/1.73 m2
* Adequate Liver Function Defined As:

  * Bilirubin (sum of conjugated + unconjugated) ≤ 1.5 x the upper limit of normal (ULN) for age
  * ALT ≤ 5 x the ULN
* Adequate Pulmonary Function Defined As: No dyspnea at rest, no exercise intolerance, and no oxygen requirement (pulse oximetry > 93% on room air).
* Adequate Cardiac Function Defined As: QTc ≤ 470 ms using Fridericia formula

Exclusion Criteria:

* CNS disease: Patients with a history of intraparenchymal CNS disease (osteosarcoma) are not eligible unless they have imaging documenting stability of CNS lesions for ≥ 3 months prior to enrollment
* Pregnancy or Breast-Feeding
* Female patients of childbearing potential are not eligible unless a negative pregnancy test result has been obtained
* Males or females of reproductive potential are not eligible unless they have agreed to use two effective methods of birth control, including a medically accepted barrier or contraceptive method
* Concomitant Medications:

  * Investigational Drugs: Subjects who are currently receiving another investigational drug are not eligible.
  * Anti-cancer Agents: Subjects who are currently receiving other anti-cancer agents are not eligible.
  * CYP3A4/5 Agents: Patients currently receiving drugs that are strong inducers or inhibitors of CYP3A4 are not eligible. Strong inducers or inhibitors of CYP3A4 should be avoided from 14 days before the 1st dose of tegavivint to the end of the study. See Appendix II for a list of agents.
  * Bisphosphonates: Patients receiving bisphosphonates within 4 Weeks of study enrollment are not eligible.
  * Denosumab: Patients who have received denosumab within 180 days prior to study enrollment are not eligible
* Infection: Subjects who have an active, uncontrolled infection.
* Subjects who have received prior solid organ or allogeneic stem cell transplantation.
* Subjects who, in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study.
* Patients with a known metabolic bone disease (ex: hyperparathyroidism, Paget's disease, osteomalacia).
* Patients with a disorder associated with abnormal bone metabolism.
* Patients with ≥ 2 grade hypocalcemia that is not corrected with oral calcium supplementation.
* Patients with vitamin D < 20 ng/mL will require supplementation or will otherwise be excluded. Patients must agree to take vitamin D +/- calcium supplements (if necessary) according to institutional or published guidelines. Additional calcium supplementation is not required if adequate dietary intake can be ascertained.
* Patients who have previously received tegavivint are not eligible.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Maximum dose tolerated | upto day 21
  The maximum tolerated dose (MTD) of Tegavivint administered intravenously over 4 hours on days 1, 8, and 15 at the dose level assigned at study entry in combination with gemcitabine. The MTD is empirically defined as the highest dose level at which no more than one patient is experiencing a dose-limiting toxicity (DLT) and the next higher dose level has been determined to be too toxic. The MTD will be determined during Cycle 1 (each cycle is 21 days)

SECONDARY OUTCOMES:
Disease control (DC) | upto 4 months
  The DC rate is defined as the number of patients without disease progression (complete response, partial response, or stable disease) during the first 4 months after enrollment
Progression-Free Survival (PFS) | End of study (upto 3 years)
  PFS will be defined as the time from enrollment to disease relapse, disease progression, or death from any cause. Patients without an event will be censored at the time of the last disease follow-up Time to event analysis of PFS will be performed using the Kaplan-Meier method
Overall Survival (OS) | End of study (upto 3 )
  Overall survival will be defined as the time from enrollment to death from any cause Time to event analysis of OS will be performed using the Kaplan-Meier method

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Cash, MD, MSc, Principal Investigator — Emory University
Locations (1):
- Arthur M. Blank Children's Healthcare of Atlanta, Atlanta, Georgia, United States